CLINICAL TRIAL: NCT04289558
Title: Safety, Feasibility, and Endothelial Effects of Sodium Nitrite Infusion in Children With Falciparum Malaria
Brief Title: Nitrite Infusion in Children With Malaria
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: current grant expiration in May, insufficient funds remaining, travel restrictions, COVID-19 restrictions in Tanzania, etc.
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100364; R01HL130763 (NIH)
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-01

CONDITIONS: Falciparum Malaria
Keywords: falciparum malaria; malaria; Africa; Duke; Tanzania; sodium nitrite; Phase I; infectious disease; hematology
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Communicable Diseases | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sodium Nitrite (Experimental): Single 60-minute intravenous infusion of sodium nitrite in 0.9% sodium chloride at up to 4 sequential dose levels (0.16, 0.32, 0.64 and 1.28 mcg/kg/minute)
  Interventions: Drug: Sodium Nitrite

INTERVENTIONS:
Drug: Sodium Nitrite — Single 60 minute infusion at 1 of 4 sequential dose levels (0.16, 0.32, 0.64 and 1.28 mcg/kg/minute). The dose amount will depend on when the participant enters the study

SUMMARY:
The purpose of this study is to assess the safety of intravenous sodium nitrite in African children who have moderately severe malaria.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study that will enroll up to 24 patients total, using a 3+3 dose escalation design, with 3 to 6 patients per dose level at up to 4 sequential dose levels (0.16, 0.32, 0.64 and 1.28 mcg/kg/minute). At each dose level patients with moderately severe malaria will receive a single 60-minute intravenous infusion of sodium nitrite in 0.9% sodium chloride. Blood pressure and methemoglobin levels will be closely monitored during the infusion and for 24 hours post infusion.

This study will allow a preliminary analysis of the safety of intravenous sodium nitrite in children with moderately severe malaria and is expected to provide preliminary data on its effects on endothelial function. The hypothesis is that sodium nitrite infusion will be safe at low dosage levels. Additionally, since deficiency of nitric oxide is linked to endothelial dysfunction in malaria, there is the hypothesis that sodium nitrite will result in improved markers of endothelial function.

Children are the largest group affected by falciparum malaria. The study population will be male children residing in Tanzania, ages 4-10 years old diagnosed with moderately severe malaria, who have been hospitalized for treatment of their malaria at Hubert Kairuki Medical University in Dar es Salaam, Tanzania. Patients will receive standard anti-malaria and supportive care treatment. The study will enroll up to 24 subjects.

Participants will receive a single intravenous infusion of sodium nitrite diluted in 0.9% sodium chloride. The infusion will be administered over 60 minutes with an infusion pump. Escala-ting doses of sodium nitrite will be administered to patients in 4 dose level cohorts. Patients will be sequentially enrolled starting at the lowest dose level. Individual patients at the same dose level will also be enrolled sequentially, such that the next patient will not receive treatment until completion of a 24- hour safety monitoring period for the prior patient. Dose assign-ment will be based on the order of study enrollment. The maximum tolerated dose (MTD) is the highest dose level wherein ≤ 1 of 6 evaluable patients experiences dose limiting toxicity (DLT). If the MTD is exceeded at the first dose level, then dosing will cease.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent from parent or legal guardian
2. Males, >4 to 10 years of age
3. Body weight > 12 kg
4. Parasitemia with Plasmodium falciparum including:

   1. Positive rapid diagnostic test result: AND
   2. >2,500 parasites/microliter by microscopy
5. Diagnosis of MSM, as follows:

   1. Clinical syndrome consistent with malaria associated with documented fever (axillary temperature >38C) or reported history of fever in the past 48 hours with no other cause present; AND
   2. Exhibiting no WHO warning signs or criteria for SM [27]
6. A negative G6PD deficiency test (careSTART G6PD quantitative biosensor)
7. Requires inpatient parenteral treatment because of inability to tolerate oral therapy
8. Hemoglobin > 8 g/dL (subjects with prior blood transfusion will be eligible).
9. Systolic blood pressure > 85 mmHg
10. Baseline quantitative methemoglobin measurement less than 2%
11. Creatinine less than the upper limit of normal

Exclusion Criteria:

1. Female gender
2. Diagnosis of severe malaria
3. Presence of infection, or mixed infection, with non-falciparum strains of malaria
4. Signs of severe malaria[27], including 1 or more of the following:

   * impaired consciousness (Blantyre coma score <3 in children)
   * prostration
   * multiple convulsions (>2 within 24 hours)
   * acidosis (base deficit >8 mEq/L or bicarbonate <15 mmol/L or lactate > 5 mmol/L)
   * hypoglycemia (blood glucose < 40 mg/dL or <2.2 mmol/L)
   * severe anemia (Hb < 5g/dL )
   * renal impairment (serum creatinine >265 uMol/L or 3 mg/dL; or blood urea >20 mmol/L)
   * jaundice (bilirubin >50 umol or 3 mg/dL with parasite count >100000/ µL)
   * pulmonary edema (including O2sat <92% with RR >30/min)
   * circulatory collapse or shock
   * significant bleeding
   * hyperparasitemia (>10%)
5. Presence of concomitant non-malarial infection
6. Known G6PD deficiency
7. Known chronic illness including renal, cardiac, pulmonary, epilepsy
8. History of a reaction to a substance or medication consisting of dyspnea and cyanosis
9. History of trauma or bleeding in the 2 weeks prior to presentation
10. Clinical impression of disseminated intravascular coagulation
11. Subjects treated with parenteral anti-malarial drugs for more than 12 hours
12. Current use of drugs with oxidative potential (e.g., nitrates, dapsone, primaquine); or drugs that cause hypotension.
13. Known allergic reactions to sodium nitrite injection

Ages: 4 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Presence of G6PD deficiency increases the risk of RBC hemolysis occurring with administration of sodium nitrite and occurrence of methemoglobinemia. G6PD deficiency is an X-linked trait, thus males are either positive or negative, while females can exhibit a range of deficiency with heterozygotes commonly having an intermediate level
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by number of subjects with at least one adverse event | 48 hours post infusion
  Adverse events will be assessed according to the NIH's Table for Grading the Severity of Adult and Pediatric Adverse Events. Events will be numerically graded 1-5; 1 being a mild event and 5 being death
Percent change in microvascular function/activation for each of the 4 dosing levels by linear regression | 48 hours post infusion
  We will assess possible covariate relationships. A model will be developed that links the pharmacokinetics with the pharmacodynamic measures of endothelial function and activation

CONTACTS AND LOCATIONS:
Locations (1):
- Hubert Kairuki Memorial University, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No